CLINICAL TRIAL: NCT03986684
Title: Targeted Analysis of Three Hormonal Systems Identifies Molecules Associated With the Presence and Severity of Nonalcoholic Fatty Liver Disease
Brief Title: Molecules Associated With the Presence and Severity of Nonalcoholic Fatty Liver Disease
Acronym: NAFLD
Status: Completed | Type: Observational
Sponsor: Hippocration General Hospital (Other)
Responsible Party: Principal Investigator, Chrysoula Boutari, Clinical Fellow, Second Propedeutic Department of Internal Medicine, MD, MSc, PhD, Hippocration General Hospital
Other Study IDs: Hippocratio_2017
Record Dates: First submitted 2019-06-07; First posted 2019-06-14 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Nonalcoholic Fatty Liver; Metabolic Syndrome
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-NAFLD
- NAFLD

SUMMARY:
Non-invasive diagnosis and treatment of nonalcoholic fatty liver disease (NAFLD) remain unmet medical needs. Aim of this study is to investigate the blood levels of three hormonal systems related to obesity, insulin resistance and inflammation in patients with different stages of NAFLD, in order to identify potential diagnostic markers.

Study aim: To compare the blood levels of: a) proglucagon-derived hormones (glucagon-like peptide [GLP]-1, GLP-2, glicentin, oxyntomodulin, glucagon, major proglucagon fragment [MPGF]), b) follistatins-activins (follistatin-like (FSTL)3, activin B), c) IGF axis (insulin-like growth factor (IGF)-1, total and intact IGF binding protein (IGFBP)-3 and IGFBP-4, in 18 individuals with early stage NAFLD vs. 14 controls To explore the levels of GDF-15, total and intact, in NAFLD versus obese controls (OC) at baseline and during oral glucose tolerance tests (OGTTs)

ELIGIBILITY:
Inclusion Criteria:

* Individuals with liver ultrasound imaging
* Adults

Exclusion Criteria:

* The presence of any secondary cause of fatty liver, such as viral, alcoholic, autoimmune and drug-induced hepatitis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects from the Second Propaedeutic Department of Internal Medicine, Ippokration Hospital, Aristotle University of Thessaloniki, Greece
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Proglucagon-derived hormones | baseline
  glucagon-like peptide GLP-1 (pg/ml)
Proglucagon-derived hormones | baseline
  glucagon-like peptide GLP-2 (pg/ml)
Proglucagon-derived hormones | baseline
  glicentin (pmol/l)
Proglucagon-derived hormones | baseline
  oxyntomodulin (pg/ml)
Proglucagon-derived hormones | baseline
  glucagon (pg/ml)
Proglucagon-derived hormones | baseline
  major proglucagon fragment [MPGF]) (ng/ml)
Follistatins-activins | baseline
  follistatin-like (FSTL)3 (ng/ml)
Follistatins-activins | baseline
  activin B (pg/ml)
IGF axis | baseline
  insulin-like growth factor (IGF)-1 (ng/ml)
IGF axis | baseline
  total and intact IGF binding protein (IGFBP)-3 and IGFBP-4 (ng/ml)
Liver ultrasound | baseline
  Estimation of echogenicity, hepatomegaly, and intra-hepatic vascular blurring (1: Intermediate, 1-2: Intermediate to Moderate, 2: Moderate, 3: Severe)
GDF-15 | baseline
  Total and intact Growth differentiation factor 15 (pg/mL)

SECONDARY OUTCOMES:
Body Mass Index (BMI) | baseline
  BMI is calculated as weight in kilograms divided by height in meters squared.
Biochemical parameters | baseline
  Glucose (mg/dl)
Biochemical parameters | baseline
  serum aspartate transaminase (AST) (U/L), ALT (U/L)
Biochemical parameters | baseline
  gamma-glutamyltransferase (GGT) (U/L)
Biochemical parameters | baseline
  total cholesterol (mg/dl), triglycerides (mg/dl) and high density lipoprotein-cholesterol (HDL-C) (mg/dl), low density lipoprotein-cholesterol (LDL-C) (mg/dl)
Biochemical parameters | baseline
  insulin (μU/ml)
Metabolomics and lipidomics analysis | baseline
  Measured with nuclear magnetic resonance spectroscopy (NMR) by Labcorp (Morrisville, USA).

CONTACTS AND LOCATIONS:
Locations (1):
- Hippokration General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boutari C, Stefanakis K, Simati S, Guatibonza-Garcia V, Valenzuela-Vallejo L, Anastasiou IA, Connelly MA, Kokkinos A, Mantzoros CS. Circulating total and H-specific GDF15 levels are elevated in subjects with MASLD but not in hyperlipidemic but otherwise metabolically healthy subjects with obesity. Cardiovasc Diabetol. 2024 May 18;23(1):174. doi: 10.1186/s12933-024-02264-5. PMID 38762719
- [Derived] Polyzos SA, Perakakis N, Boutari C, Kountouras J, Ghaly W, Anastasilakis AD, Karagiannis A, Mantzoros CS. Targeted Analysis of Three Hormonal Systems Identifies Molecules Associated with the Presence and Severity of NAFLD. J Clin Endocrinol Metab. 2020 Mar 1;105(3):e390-400. doi: 10.1210/clinem/dgz172. PMID 31690932